CLINICAL TRIAL: NCT02129790
Title: Mentalization-Based Therapy to Prevent Suicidal Behavior in Adolescents With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-000988
Record Dates: First submitted 2014-04-25; First posted 2014-05-02 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Bipolar Disorder; Suicidal Ideation
Keywords: Bipolar Disorder; Suicidal; Depression; Self-harm; Psychosocial intervention
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation; Depression; Self-Injurious Behavior | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mentalization-Based Therapy (Experimental): Up to 21 individual MBT-A sessions plus 9 monthly family sessions. MBT-A will include psychoeducation and coping strategies.
  Interventions: Behavioral: Mentalization-Based Therapy

INTERVENTIONS:
Behavioral: Mentalization-Based Therapy — Up to 21 individual MBT-A sessions plus 9 monthly family sessions. MBT-A sessions will focus on the adolescent's recent social experiences and the resulting mental states and managing interpersonal challenges, particularly those involving separation or loss. The goal of this intervention is to improve the adolescent's ability to mentalize: to understand, acknowledge, and predict thoughts and feelings in oneself and others.

SUMMARY:
Children and adolescents with early-onset bipolar disorder (BD) are at high risk for intentionally hurting themselves. Although there are therapies in existence for these youths with BD, they do not address suicide prevention specifically. Mentalization-based therapy for adolescents (MBT-A) has been shown to be helpful in reducing self-harm in the adolescent and adult population with borderline personality disorder. The investigators will modify the MBT-A treatment procedures for persons with BD who have had a recent period of suicidal ideation or behavior.

DETAILED DESCRIPTION:
Youth with early-onset bipolar disorder (BD) are at an elevated risk for intentional self-harm compared to healthy adolescents or adolescents with other psychiatric disorders. Adolescents vulnerable to emotion dysregulation and self-harm often have deficits in the ability to mentalize: to understand, acknowledge, and predict thoughts and feelings in oneself and others. Mentalization-based therapy for adolescents (MBT-A) has been shown to be more effective than 'usual care' in reducing self-harm for adolescents and adults with borderline personality disorder. MBT-A includes psychoeducational and coping strategies that may prove quite effective for bipolar adolescents who are at elevated risk for self-harm.

Participation in this study will last 9 months. All participants will receive a thorough medical-psychiatric evaluation. All youth will be able to receive pharmacotherapy with a study psychiatrist in the CHAMP clinic. The MBT-A will consist of up to 21 weekly, biweekly and monthly individual sessions interspersed with 9 monthly family sessions (30 therapy hours total). Participants will also complete follow-up assessments every 3 months for 9 months. These assessments will include research interviews and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Bipolar Disorder I, Bipolar Disorder II, or Bipolar Disorder Not Otherwise Specified
* Living with or in close contact with at least one parent who is willing to participate
* Have had at least 1 week in the prior 3 months of significant suicidal ideation and/or at least one suicidal event in the 3 months prior to study intake.
* Willing to be treated pharmacologically by a psychiatrist in the UCLA Child and Adolescent Mood Disorders (CHAMP) clinic

Exclusion Criteria:

* Participants requiring immediate hospitalization
* Diagnosis of borderline personality disorder, schizophrenia, or schizoaffective disorder.
* Current substance dependence disorder

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Self-harm Scores | measured every 3 months for 9 months
  Self-harm is a composite score derived from two Kiddie Schedule for Affective Disorders and Schizophrenia Depression Rating Scale items, total scores on the Harkavy-Asnis Suicide Scale, total scores on the Risk and Self-Harm Scale, and specific levels of ideation or behavior on the Columbia Suicide and Self-Harm Scale.

SECONDARY OUTCOMES:
Treatment completion | first 6 study months
  Treatment completion will be measured by number of sessions attended and number of patients who drop out of treatment before six months.
Depression scores | every 3 months for 9 months
  Depression is a total score drawn from the Kiddie Schedule for Affective Disorders and Schizophrenia, Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: David J Miklowitz, Ph.D., Principal Investigator — UCLA Department of Psychiatry
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Miklowitz DJ, Taylor DO. Family-focused treatment of the suicidal bipolar patient. Bipolar Disord. 2006 Oct;8(5 Pt 2):640-51. doi: 10.1111/j.1399-5618.2006.00320.x. PMID 17042836
- [Background] Rossouw TI, Fonagy P. Mentalization-based treatment for self-harm in adolescents: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Dec;51(12):1304-1313.e3. doi: 10.1016/j.jaac.2012.09.018. PMID 23200287
- See also: UCLA Child and Adolescent Mood Disorders Program — http://www.semel.ucla.edu/champ